CLINICAL TRIAL: NCT00541736
Title: Glyceryl-Trinitrate-Induced Headache in Patients With Familial Hemiplegic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Collaborators: EUROHEAD (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FHM-GTN-2007-08
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Familial Hemiplegic Migraine
Keywords: Familial Hemiplegic Migraine
MeSH Terms: conditions — Migraine with Aura | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): GTN-infusion
  Interventions: Drug: Nitroglycerine
- Controls (Active Comparator): GTN-infusion
  Interventions: Drug: Nitroglycerine

INTERVENTIONS:
Drug: Nitroglycerine — Nitroglycerine infusion over 20 minutes: 0.5 ug/kg/min

SUMMARY:
The aim of the present study is to explore the importance of migraine genes on the headache/migraine responses after GTN in FHM-patients and healthy volunteers.

DETAILED DESCRIPTION:
Glyceryl trinitrate (GTN) induces migraine attacks indistinguishable from spontaneous attacks in approximately 80% of migraine sufferers. After systemic administration GTN is transformed to nitric oxide (NO). Treatment of spontaneous migraine attacks with an inhibitor of NO is effective in 60% of patients. These data show that NO is involved in both initiation and maintenance of migraine attack.

The importance of migraine genes is disputed. Evidence from FHM patients with known mutations indicates that migraine pathways in FHM may be different from normal migraine. The aim of the present study is to examine whether this difference also exists in FHM patients without known mutations. The project will improve our understanding of the neurobiology of migraine and stimulate development of new treatment targets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of familial hemiplegic migraine (IHS-classification criteria)

Exclusion Criteria:

Patients and controls:

* A history of cerebrovascular disease and other CNS- disease
* A history of serious somatic and mental disease
* A history suggesting ischaemic heart disease
* A history of hypo- or hypertension
* Daily intake of medication apart from oral contraceptives
* Abuse of alcohol or medicine (opioid analgesics).
* Pregnant or breastfeeding women.

On the study day:

* No intake of a simple analgesic in the previous 48 hours
* No headache in the previous 48 hours

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Migraine and associated symptoms | 0-14 h
Migraine aura | 0 - 14 h

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Møller Hansen, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, University of Copenhagen, Faculty of Health Sciences, Department of Neurology, Glostrup Hospital, Glostrup, Copenhagen, Denmark